CLINICAL TRIAL: NCT01055483
Title: A Phase Ib, Open-label, Multi-center Dose-finding Study of Oral Panobinostat (LBH589) in Combination With Ara-C and Mitoxantrone as Salvage Therapy for Refractory or Relapsed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B2116; 2008-002986-30 (EudraCT Number)
Record Dates: First submitted 2010-01-21; First posted 2010-01-25 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2013-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; AML; relapsed acute myeloid leukemia; refractory acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Panobinostat

ARMS (1):
- LBH589 (Experimental)
  Interventions: Drug: panobinostat/LBH589B

INTERVENTIONS:
Drug: panobinostat/LBH589B

SUMMARY:
The study will determine the maximal tolerated dose (MTD) of panobinostat administered in combination with a fixed combination of cytarabine (ara-C) and mitoxantrone in adult patients with relapsed or refractory acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Patients with cytopathologically confirmed diagnosis of AML according to WHO criteria, excluding acute promyelocytic leukemia.
* First relapsed AML
* Primary refractory AML defined as failure to respond to initial induction chemotherapy (no CR) or recurrence within 6 months of initial CR.
* Age more than 18 years
* ECOG performance status < 2

Exclusion Criteria:

* Prior treatment with deacetylase inhibitor
* Concurrent therapy with any other investigational agent
* Patients who have received cumulative doses (or its equivalent to other anthracyclines) of more than 360 mg/m2 of doxorubicin will be excluded from the study.
* Clinical symptoms suggesting CNS leukemia
* LVEF below 45% Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) | 1 cycle (1 cycle = 28 days)

SECONDARY OUTCOMES:
Frequency, severity and duration of Adverse Events (AE) using CTCAE version 3.0 | During maximal three LBH589/chemotherapy cycles and subsequent optional single-agent LBH589 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Novartis Investigative Site, Paris, France
- Germany (4):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Ulm

REFERENCES:
- See also: Results for LBH589B2116 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=8103